CLINICAL TRIAL: NCT02280538
Title: A Randomized Placebo Controlled Trial to Assess the Structural Effect and Long-term Symptomatic Relief of Repeated Intra-articular Injections of Hyaluronic Acid in Primary Knee Osteoarthritis
Brief Title: Trial to Assess the Structural Effect and Long-term Symptomatic Relief of Intra-articular Injections of Hyaluronic Acid in Primary Knee OA
Acronym: ViscOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: NOVA Medical School (Other); Centro de Estudos de Doenças Crónicas (Other); Hospital de Santa Maria, Portugal (Other); Hospital de Egas Moniz (Other); Instituto de Medicina Molecular João Lobo Antunes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOVA-FCM-Rheuma-2
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis Of Knee
Keywords: Knee Osteoarthritis; Intra-Articular Hyaluronic Acid; disease modifying
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-Articular Hyaluronic Acid (Experimental): hylan G-F 20 (high molecular weight hyaluronic acid):
  * intra-articular administration
  * 6 mL
  * administered every 6 months
  * for 2 years
  Interventions: Device: Intra-Articular Hyaluronic Acid
- Placebo (Placebo Comparator): Saline solution:
  * intra-articular administration
  * 6 mL
  * administered every 6 months
  * for 2 years
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Intra-Articular Hyaluronic Acid
  Other Names: hylan GF-20
  Arms: Intra-Articular Hyaluronic Acid
Device: Placebo
  Arms: Placebo

SUMMARY:
The present study is designed to test the hypothesis that Intra-Articular Hyaluronic Acid (IAHA) is superior to placebo in slowing structural progression and on long term symptomatic effect in primary knee Osteoarthritis (OA) patients.

The investigators will perform a multicenter double-blind, randomized, placebo-controlled, parallel group trial.

DETAILED DESCRIPTION:
The target population will be patients with the diagnosis of knee osteoarthritis who are followed at two Portuguese hospitals (Centro Hospitalar de Lisboa Norte - Hospital Santa Maria, Centro Hospitalar de Lisboa Ocidental - Hospital Egas Moniz).

All patients selected will be included in the intention-to-treat group. Then, using blocked randomization method they will be assigned to receive either IAHA, or placebo (saline solution). At both hospitals the study will consist of four injections of IAHA, 6 months apart, plus a 6 month period after the injection, resulting in a total follow-up period of 24 months. Before each new cycle a follow-up consultation will be performed in order to assess pain and function (KOOS), quality of life (SF-36), adverse events and consumption of acetaminophen and NSAIDS regarding the week before evaluation. X-rays will be performed in the beginning of follow-up, one year after that and 6 months after the last cycle of IAHA or placebo injections (24 months).

Ultrasound evaluation will be performed at the target knee in same time points as X-rays by two rheumatologists trained in musculoskeletal ultrasound examination. Additionally, the investigators will assess potential biochemical biomarkers of knee OA structural progression and response to treatment. Measurements will be performed in both serum and urine and, If possible, synovial fluid aspiration will be performed and together with blood and urine samples stored at the Biobanco-IMM Instituto de Medicina Molecular for analysis. Biologic samples collection will be performed at baseline and repeated at the 4th, 12th, 24th, 36th weeks, and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee OA as defined by the ACR clinical and radiographic criteria
* Kellgren-Lawrence grade of II or III on prior x-rays (taken within 6 months of the screen visit) or screen X-ray
* A minimum medial and/or lateral JSW of the target knee of 2 mm
* Knee pain of 40 mm or greater on a 100 mm visual analogue scale (VAS) at any time during the week before inclusion
* Oral corticosteroids (≤10 mg/day prednisolone or equivalent), NSAIDs, and acetaminophen are permitted if the dose had been stable for at least one month prior to baseline

Exclusion Criteria:

* Body mass index greater than 40 kg/m2
* Varus or valgus deformity of the knee > 15 degrees (assessed by goniometry)
* History of trauma, surgery or planned surgery to the study joint (including arthroscopy surgery), joint inflammatory diseases, septic arthritis and/or microcrystalline arthropathies
* Coagulation/platelet disorders
* Active malignancy, active systemic infection, or any contraindication to MRI
* Potent analgesics including opiates, oral corticosteroid therapy within one month prior to enrolment into the study other than stable doses of ≤ 10 mg daily prednisolone or equivalent
* Knee administration of intra-articular steroids in the previous 3 months or HA injections during the past year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Joint Space Width | 2 years
  Mean change of minimal JSW of the most affected compartment of the tibiofemural joint in both placebo and IAHA groups at the end of follow-up (2 years).

SECONDARY OUTCOMES:
OMERACT/OARSI 2004 response | 6 months
  Proportion of patients achieving symptomatic relief according to OMERACT/OARSI 2004 response criteria at 6 months of follow-up in both placebo and IAHA groups. OMERACT/OARSI 2004 will be determined using KOOS questionnaire.
OMERACT/OARSI 2004 response | 2 years
  Proportion of patients achieving symptomatic relief according to OMERACT/OARSI 2004 criteria at each follow-up visit. OMERACT/OARSI 2004 will be determined using KOOS questionnaire.
Ocurrence of Knee replacement surgery | 2 years
  Proportion of patients submitted to knee replacement surgery at the end of follow-up
Acetaminophen Consumption | 2 years
  Mean consumption of acetaminophen (mg/day) at each follow-up visit.
NSAIDs | 2 years
  Mean consumption of NSAIDs (mg/day) at each follow-up visit.
SF-36 questionnaire - Physical Score | 2 years
  Mean score of SF-36 questionnaire at each follow-up visit.
SF-36 questionnaire - Mental Score | 2 years
  Mean score of SF-36 questionnaire at each follow-up visit.
Euro QoL 5D | 2 years
  Mean score of Euro QoL 5D questionnaire at each follow-up visit.
Adverse events | 2 years
  Total number of adverse events occurring on both placebo and IAHA groups at each follow-up visit.
Visual Analog Scale | 2 years
  Mean VAS score at 2 years
Visual Analog Scale | 2 years
  Mean VAS score at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime C Branco, MD, PhD, Principal Investigator — CEDOC; Alexandre Sepriano, MD, Study Director — Centro Hospitalar de Lisboa Ocidental; João Gomes, MD, Study Chair — Centro Hospitalar de Lisboa Ocidental
Locations (2):
- Portugal (2):
  - Centro Hospitalar de Lisboa Ocidental - Hospital Egas Moniz, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Norte, Lisbon